CLINICAL TRIAL: NCT03103152
Title: PROVENT: A Randomised, Double Blind, Placebo Controlled Feasibility Study to Examine the Clinical Effectiveness of Aspirin and/or Vitamin D3 to Prevent Disease Progression in Men on Active Surveillance for Prostate Cancer
Brief Title: A Study to Examine the Effectiveness of Aspirin and/or Vitamin D3 to Prevent Prostate Cancer Progression
Acronym: PROVENT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: Barts and the London School of Medicine and Dentistry (Other); Cancer Research UK (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: isrctn91422391
Record Dates: First submitted 2016-11-21; First posted 2017-04-06 (Actual); Results first posted 2023-03-29 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2020-03

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Active Surveillance; Chemo-prevention
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Aspirin; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- High dose Aspirin & Vitamin D (Experimental): Aspirin high dose (300mgs) daily & Vitamin D 4,000 IU (0.1mg) per day
  Interventions: Drug: High dose Aspirin & Vitamin D
- High dose Aspirin, Vitamin D placebo (Experimental): high dose aspirin (300mgs) daily and Vitamin D placebo (Miglyol®812 Oil)
  Interventions: Drug: High dose Aspirin, Vitamin D placebo; Drug: Aspirin placebo, Vitamin D placebo
- Low dose Aspirin , Vitamin D (Experimental): Low dose aspirin (100mgs) daily & Vitamin D 4,000 IU (0.1mg) per day
  Interventions: Drug: Low dose Aspirin , Vitamin D
- Low dose Aspirin, Vitamin D placebo (Placebo Comparator): Low dose aspirin (100mgs) daily and Vitamin D placebo (Miglyol®812 Oil)
  Interventions: Drug: Low dose Aspirin, Vitamin D placebo
- Aspirin Placebo, Vitamin D (Experimental): Aspirin placebo and Vitamin D active ingredient - Vigantol® Oil
  Interventions: Drug: Low dose Aspirin , Vitamin D; Drug: Aspirin Placebo, Vitamin D
- Aspirin placebo, Vitamin D placebo (Experimental): Aspirin placebo and Vitamin D placebo - Miglyol®812 Oil
  Interventions: Drug: Aspirin placebo, Vitamin D placebo

INTERVENTIONS:
Drug: High dose Aspirin & Vitamin D — Aspirin 1 x 300mg tablet daily & Vitamin D 4,000IU daily. (8 drops).
  Other Names: Aspirin - acetylsalicylic acid; Vitamin D - Vigantol® Oil
  Arms: High dose Aspirin & Vitamin D
Drug: High dose Aspirin, Vitamin D placebo — Aspirin 1 x 300mg tablet daily & Vitamin D placebo (8 drops).
  Other Names: Aspirin - acetylsalicylic acid; Vitamin D placebo - Miglyol®812 Oil
  Arms: High dose Aspirin, Vitamin D placebo
Drug: Low dose Aspirin , Vitamin D — Aspirin 1 x 100mg tablet daily & Vitamin D 4,000IU daily. (8 drops).
  Other Names: Aspirin - acetylsalicylic acid; Vitamin D - Vigantol® Oil
  Arms: Aspirin Placebo, Vitamin D; Low dose Aspirin , Vitamin D
Drug: Low dose Aspirin, Vitamin D placebo — Aspirin 1 x 100mg tablet daily & Vitamin D placebo 8 drops daily.
  Other Names: Aspirin - acetylsalicylic acid; Vitamin D placebo - Miglyol®812 Oil
  Arms: Low dose Aspirin, Vitamin D placebo
Drug: Aspirin Placebo, Vitamin D — Aspirin 1 x 300mg placebo tablet daily & Vitamin D 4,000IU daily. (8 drops).
  Other Names: Vitamin D - Vigantol® Oil
  Arms: Aspirin Placebo, Vitamin D
Drug: Aspirin placebo, Vitamin D placebo — Aspirin 1 x 100mg placebo tablet daily & Vitamin D 4,000IU daily. (8 drops).
  Other Names: Aspirin Placebo, Vitamin D; Vitamin D placebo - Miglyol®812 Oil
  Arms: Aspirin placebo, Vitamin D placebo; High dose Aspirin, Vitamin D placebo

SUMMARY:
To demonstrate the acceptability and feasibility of recruitment to a randomised chemoprevention study of standard (300mg) or low dose (100mg) aspirin vs. placebo and/or Vitamin D3 vs. placebo in patients enrolled on an Active Surveillance programme for prostate cancer.

DETAILED DESCRIPTION:
The PROVENT study is a randomised, double blind, placebo controlled feasibility study to examine the clinical effectiveness of aspirin and/or Vitamin D3 to prevent disease progression in men on Active Surveillance for prostate cancer

The main outcome measure of the trial is the rate of patient recruitment to a randomised chemoprevention study in men enrolled on an Active Surveillance programme for prostate cancer

Secondary outcomes include the response to treatment as determined by serial multi-parametric magnetic resonance imaging (MRI) of the prostate, biochemical disease progression and histological disease progression after 12 months of therapy and finally toxicity and/or allergy to both aspirin and Vitamin D3.

ELIGIBILITY:
1. Male subjects aged 16 years or over with an estimated life expectancy of more than three years
2. Willing and able to provide written informed consent
3. Corrected serum calcium ≤ 2.65mmol/l
4. No previous treatment for prostate cancer (including surgery, hormone therapy, radiotherapy, cryotherapy)
5. Must have undergone a multi-parametric MRI of the prostate, deemed assessable by the local radiologist, and any lesions seen must have undergone targeted biopsy, (transrectal or transperineal) within 12 months of study registration.
6. Histologically confirmed prostate cancer* following prostate biopsy (including at least 10 cores of prostate tissue) in men opting for Active Surveillance as their primary cancer therapy.

   * PROVENT Prostate Cancer Criteria. All must be met for Inclusion:

     * Gleason score 6 or 7 (Gleason 3+3 or 3+4)
     * Clinical and radiological stage <T3
     * Serum Prostate Specific Antigen (PSA) ≤15.0 ng/ml
     * Less than 10mm of cancer in a single core

Exclusion Criteria:

1. Previously treated prostate cancer (including radiotherapy, hormone therapy, brachytherapy or surgery)
2. Currently enrolled, or has been a participant within the last 30 days, in any other investigational drug or device study.
3. Current daily use of aspirin or NSAIDs; or daily dietary supplements/medication containing more than 400 IU (10 micrograms per day) Vitamin D; or chronic use (defined as > 6 months continuous daily use) of either aspirin or >400IU Vitamin D within two years of study enrolment
4. Current or previous use of 5-α reductase inhibitors such as finasteride or dutasteride
5. Not willing to comply with the procedural requirements of this protocol including repeat prostate biopsies
6. Known allergy/sensitivity to or intolerance of aspirin, other salicylates or NSAIDs e.g. ibuprofen/ naproxen
7. Prior history of gastro-intestinal bleeding or ulceration, severe dyspepsia or inflammatory bowel disease
8. Haemophilia or other bleeding diatheses
9. Prior history of renal stone disease
10. Chronic renal disease (≥stage 4)
11. Known hypercalcaemia (corrected serum calcium >2.65 mmol/l) or untreated hyperparathyroidism
12. Any bowel condition that would make repeat transrectal biopsy hazardous or difficult to perform e.g. recto-urethral fistula, or prior bowel surgery such as abdomino-perineal resection.
13. Any malignancy (other than non-melanoma skin cancer) that has not been in complete remission for five years
14. Any serious co-existent medical condition that would make repeat prostate biopsy hazardous e.g. anti-coagulation requiring continuous administration
15. Severe Asthma
16. G6PD ( glucose-6-phosphate dehydrogenase) deficiency
17. Pre-existing macular degeneration
18. All contraindications to aspirin and Vitamin D3 (e.g. Sarcoidosis), including concomitant therapy with any medication that may interact with aspirin or Vitamin D3 (see section 4.10)
19. Tuberculosis
20. Regular consumption of alcohol units greater than the recommended daily limit of 3-4 units per day (men)

Ages: 16 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2016-12; Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Greg Shaw, MD, Principal Investigator — Queen Mary London; Jack Cuzick, PhD, Study Director — Queen Mary London
Locations (7):
- United Kingdom (7):
  - Darent Valley Hospital, Dartford
  - University Hospital of Wales, London
  - University Hospital UHCW NHS Trust, London
  - St Bartholomews Hospital London, Bart's and the London school of Medicine, London
  - University College Hospital London, London
  - Homerton Hospital, London
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 12 months recruitment (December 2016 to Dec 2017). All recruitment took place in the hospital setting within active surveillance clinics.
Pre-assignment Details: Helicobacter pylori (H. pylori) has been shown to be a causative factor in GI bleeding, so all participants were tested for this at randomisation as a precaution. Patients who tested positive were prescribed a course of proton pump inhibitors(PPIs) & antibiotics if they wished to continue on the study. GPs were informed. Serum calcium levels were also checked at baseline. Anyone with symptoms of hypercalcaemia was excluded.
Period: Overall Study
Arm/Group | High Dose Aspirin & Vitamin D | High Dose Aspirin, Vitamin D Placebo | Low Dose Aspirin , Vitamin D | Low Dose Aspirin, Vitamin D Placebo | Aspirin Placebo, Vitamin D | Aspirin Placebo, Vitamin D Placebo
Started | 17 | 16 | 19 | 18 | 16 | 18
Completed | 7 | 10 | 8 | 9 | 10 | 9
Not Completed | 10 | 6 | 11 | 9 | 6 | 9
Not completed — Physician Decision | 5 | 2 | 6 | 3 | 3 | 1
Not completed — Protocol Violation | 2 | 2 | 1 | 2 | 1 | 1
Not completed — Inter-current illness | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 1 | 1 | 1
Not completed — Patient wishes to come off active surveillance | 2 | 0 | 1 | 1 | 1 | 3
Not completed — Unacceptable side effects | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 1 | 0 | 1
Not completed — Testicular pain | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose Aspirin & Vitamin D | High Dose Aspirin, Vitamin D Placebo | Low Dose Aspirin , Vitamin D | Low Dose Aspirin, Vitamin D Placebo | Aspirin Placebo, Vitamin D | Aspirin Placebo, Vitamin D Placebo | Total
Number analyzed (Participants) | 17 | 16 | 19 | 18 | 16 | 18 | 104
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 56 [54 to 64] | 61 [55.75 to 64.5] | 62 [60 to 68.5] | 59.5 [56 to 65.75] | 64 [56.75 to 66] | 65.5 [57 to 70.75] | 61 [56 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 17 | 16 | 19 | 18 | 16 | 18 | 104
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Rate of Patient Recruitment to a Randomised Chemoprevention Study in Men Enrolled on an Active Surveillance Programme for Prostate Cancer. Number Accrued Per Month.
Description: The proportion of eligible patients that join the trial over the 12-month trial recruitment period.
Time Frame: 12 months
Population: Number accrued by arm over the 12 month recruitment period.
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose Aspirin & Vitamin D | High Dose Aspirin, Vitamin D Placebo | Low Dose Aspirin , Vitamin D | Low Dose Aspirin, Vitamin D Placebo | Aspirin Placebo, Vitamin D | Aspirin Placebo, Vitamin D Placebo
Number analyzed (Participants) | 17 | 16 | 19 | 18 | 16 | 18
Participants | 17 | 16 | 19 | 18 | 16 | 18

2. Secondary Outcome: Response to Treatment as Determined by Serial Multi-parametric Magnetic Resonance Imaging (MRI) of the Prostate. New Lesion Present or Existing Lesion + or - in Size.
Description: Radiological progression was defined as 'development of a Prostate Imaging-Reporting and Data System (PI-RADS) 4/5 lesion (17) on mpMRI, where no lesion was identified before, 33% volume increase in the size of the lesion, or radiological upstaging to T3 or above based on local site reports.' Absence of these features represented radiologically stable disease.
  Lesion on multi-parametric imaging where no MRI lesion at screening. An MRI scan shows a screening + or - in volume by > 33%, or an upgrading of MRI stage of disease to ≥3.
Time Frame: 3 years
Population: All participants with a baseline & 12 mth MRI scan.
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose Aspirin & Vitamin D | High Dose Aspirin, Vitamin D Placebo | Low Dose Aspirin , Vitamin D | Low Dose Aspirin, Vitamin D Placebo | Aspirin Placebo, Vitamin D | Aspirin Placebo, Vitamin D Placebo
Number analyzed (Participants) | 9 | 8 | 8 | 5 | 9 | 8
Participants
  Disease Regression | 1 | 5 | 5 | 0 | 3 | 2
  Stable Disease | 4 | 3 | 2 | 4 | 6 | 6
  Disease Progression | 4 | 0 | 1 | 1 | 0 | 0

3. Secondary Outcome: Number of Participants With Biochemical (PSA) Disease Progression
Description: 50% increase in serum Prostate Specific Antigen at 12 months from baseline.
Time Frame: 12 months
Population: Number of subjects analysed
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose Aspirin & Vitamin D | High Dose Aspirin, Vitamin D Placebo | Low Dose Aspirin , Vitamin D | Low Dose Aspirin, Vitamin D Placebo | Aspirin Placebo, Vitamin D | Aspirin Placebo, Vitamin D Placebo
Number analyzed (Participants) | 12 | 13 | 11 | 10 | 12 | 15
Participants
  Disease Regression | 1 | 2 | 0 | 0 | 0 | 1
  Stable Disease | 9 | 10 | 10 | 10 | 10 | 13
  Disease Progression | 2 | 1 | 1 | 0 | 2 | 1

4. Secondary Outcome: Number of Participants With Histological Disease Progression
Description: Histological disease progression will be defined as an increase in Gleason scores from: Gleason 3+3 to Gleason score 7 or higher Gleason 3+4 (score 7) to 4+3 (score 7) or Gleason 4+3 to a higher score
  Or a 50% increase in maximum cancer core length (MCCL)
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose Aspirin & Vitamin D | High Dose Aspirin, Vitamin D Placebo | Low Dose Aspirin , Vitamin D | Low Dose Aspirin, Vitamin D Placebo | Aspirin Placebo, Vitamin D | Aspirin Placebo, Vitamin D Placebo
Number analyzed (Participants) | 17 | 16 | 19 | 18 | 16 | 18
Participants | 2 | 7 | 5 | 2 | 3 | 6

5. Secondary Outcome: Number of Patients With Adverse With Toxicity, Allergy or Symptoms From Aspirin or Vitamin D
Description: Aspirin toxicity: Haemorrhagic stroke, anaphylaxis following administration, gastrointestinal bleeding requiring intervention (both medical and surgical)
  Vitamin D3 toxicity: Hypercalcaemia, Anaphylaxis
Time Frame: 18 months + 30 days
Population: Total intention to treat population.
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose Aspirin & Vitamin D | High Dose Aspirin, Vitamin D Placebo | Low Dose Aspirin , Vitamin D | Low Dose Aspirin, Vitamin D Placebo | Aspirin Placebo, Vitamin D | Aspirin Placebo, Vitamin D Placebo
Number analyzed (Participants) | 17 | 16 | 19 | 18 | 16 | 18
Participants
  Haemorrhagic Stroke | 0 | 0 | 0 | 0 | 0 | 1
  Rectal Bleeding | 0 | 0 | 2 | 0 | 0 | 0
  Anaphylaxis either Vit D or Aspirin | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcaemia | 0 | 0 | 0 | 0 | 0 | 0
  None of the above toxicities | 17 | 16 | 17 | 18 | 16 | 17

ADVERSE EVENTS:
Time Frame: Adverse events were monitored/assessed from the date of first randomisation (in December 2016) until the end of the trial (June 2018) +30 day pharmacovigilance period Overall: AEs reported from the date of each patient's randomisation until their last visit within 18 months after randomisation + 30 days pharmacovigilance. Per patient: participants were followed from the point of recruitment until 18 months after recruitment for each participant +30 days for pharmacovigilance.
Description: Since there is no risk arising from the transfer of any PROVENT IMP products via seminal fluid, it has been deemed unnecessary to collect & record pregnancies where the father is a PROVENT study participant.
  Mild: Some discomfort noted but without disruption of daily life Moderate: Discomfort enough to affect/reduce normal activity Severe: Complete inability to perform daily activities and lead a normal life Unknown. Intensity not be confused with regulatory definition "serious".
Arm/Group | High Dose Aspirin & Vitamin D | High Dose Aspirin, Vitamin D Placebo | Low Dose Aspirin , Vitamin D | Low Dose Aspirin, Vitamin D Placebo | Aspirin Placebo, Vitamin D | Aspirin Placebo, Vitamin D Placebo
All-Cause Mortality (participants affected / at risk) | 0/17 | 1/16 | 0/19 | 0/18 | 0/16 | 0/18
Serious Adverse Events (participants affected / at risk) | 2/17 | 2/16 | 2/19 | 1/18 | 1/16 | 0/18
Other Adverse Events (participants affected / at risk) | 5/17 | 9/16 | 6/19 | 4/18 | 7/16 | 11/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose Aspirin & Vitamin D (N=17) | High Dose Aspirin, Vitamin D Placebo (N=16) | Low Dose Aspirin , Vitamin D (N=19) | Low Dose Aspirin, Vitamin D Placebo (N=18) | Aspirin Placebo, Vitamin D (N=16) | Aspirin Placebo, Vitamin D Placebo (N=18)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mass in brain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary Retention Post-operative (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile Infection (Infections and infestations) | 0 | 1 | 1 | 0 (0) | 0 (0) | 0 (0)
Testicular Pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 (1) | 0 (0) | 0 (0)
Rectal Bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose Aspirin & Vitamin D (N=17) | High Dose Aspirin, Vitamin D Placebo (N=16) | Low Dose Aspirin , Vitamin D (N=19) | Low Dose Aspirin, Vitamin D Placebo (N=18) | Aspirin Placebo, Vitamin D (N=16) | Aspirin Placebo, Vitamin D Placebo (N=18)
Abdominal aortic aneurysm (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal crampy pains (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acid Reflux (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute Back Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arm Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood in urine (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Pressure Increased (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood in stool (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest Infection (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coccyx Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cold (General disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fast Heart Beat (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fractured Ribs (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemospermia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hay Fever (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head Cold (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Indigestion (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Mouth Ulceration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nose Bleed (General disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Stomach Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prolapsing Haemorrhoid (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal Bleeding (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sore Throat (General disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomach Acid (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Swelling Right Testicle (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swollen Toes (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower urinary tract symptoms (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nocturia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary Retention (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Back Ache (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacterial Infection (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) — Helicobacter pylori
Bleeding Post-op (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dark Circles Under Eyes (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flu-like symptoms (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flu Prophylaxis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Left Hip Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Left Knee Meniscal Tear (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leg Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lichen Simplex (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in hips, knees, shoulders (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pins & Needles (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Polymyalgia Rheumatica (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post-op Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash, headache, insomnia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Removal of basal cell (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomach Ache (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upset Stomach (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary Urgency (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post procedural constipation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Teary Eyes (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear Infection (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal relux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary Incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fever (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The NHS Organisation shall not publish/disseminate the conclusions of the Study, including all or any part of the Results of the Study without the prior written consent of the Sponsor. Any publication/dissemination of the conclusions of the Study by the NHS Organisation shall not occur until the Sponsor has published the conclusions of the Study in accordance with clause 7.2 and shall refer to publication by the Sponsor in such form as the Sponsor may reasonably direct.

DOCUMENTS (2):
  • Study Protocol (2019-10-28): https://cdn.clinicaltrials.gov/large-docs/52/NCT03103152/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-17): https://cdn.clinicaltrials.gov/large-docs/52/NCT03103152/SAP_001.pdf